CLINICAL TRIAL: NCT06219928
Title: Comparison of the Effects of Dexmedetomidine and Ketamine Infusion on the Inflammatory Response in Liver Resection: a Randomized Double-blind Placebo Study
Brief Title: Comparison of the Effects of Dexmedetomidine and Ketamine Infusion on the Inflammatory Response in Liver Resection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, irem ateş, Associate Professor as the Principal Investigator, Ataturk University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: B.30.2.ATA.0.01.OO/6
Record Dates: First submitted 2024-01-03; First posted 2024-01-23 (Actual); Last update posted 2024-11-18 (Actual); Status verified 2024-11

CONDITIONS: Inflammation; Analgesia
Keywords: Liver resection; ketamine; dexmedetomidine; inflammation
MeSH Terms: conditions — Inflammation; Agnosia | interventions — Control Groups; Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Saline (Active Comparator): After intubation, saline infusion will be started. The control group will also be infused with the same volume of saline..
  Interventions: Procedure: Control Group
- Ketamine (Active Comparator): After intubation, the patient will be started on ketamine infusion at a low dose of 0.25mg/kg/hour.
  Interventions: Procedure: Ketamine Group
- Dexmedetomidine (Active Comparator): After intubation, the patient will be infused at a low dose of 1 mg/kg dexmedetomidine for the first 10 minutes, then 0.5 mg/kg/hour
  Interventions: Procedure: Dexmedetomidine

INTERVENTIONS:
Procedure: Control Group — After intubation, saline infusion will be started. The control group will also be infused with the same volume of saline
  Arms: Saline
Procedure: Ketamine Group — After intubation, the patient will be started on ketamine infusion at a low dose of 0.25mg/kg/hour.
  Arms: Ketamine
Procedure: Dexmedetomidine — After intubation, the patient will be infused at a low dose of 1 mg/kg for the first 10 minutes, then 0.5 mg/kg/hour.
  Arms: Dexmedetomidine

SUMMARY:
Resection is being performed with increasing frequency in the treatment of surgical diseases of the liver. Ischemia-reperfusion injury is a major cause of liver injury occurring during surgical procedures, including hepatic resection and liver transplantation. Dexmedetomidine and ketamine, which are frequently used in anesthesia practice, also have strong anti-inflammatory capacity. The primary aim of this study is to investigate the effect of iv low-dose ketamine and dexmedetomidine infusion on inflammation in liver resection surgery, and the secondary aim is to determine its effect on pain scores.

DETAILED DESCRIPTION:
General anesthesia will apply to all patients. Group 1 (Control Group, n=15); After intubation, saline infusion will be started. The control group will also be infused with the same volume of saline.

Group 2 (Ketamine Group, n=15); After intubation, the patient will be started on ketamine infusion at a low dose of 0.25mg/kg/hour.

Group 3 (Dexmedetomidine Group, n=15); After intubation, the patient will be infused at a low dose of 1 mg/kg for the first 10 minutes, then 0.5 mg/kg/hour.

For biochemical examination, blood will be taken for PEDF (Pigment epithelium-derived factor), Pentraxin 3, Serum amyloid A at the 1st and 12th postoperative hour. AST, ALT, GGT, LDH, bilirubin, CRP and hemogram results, which are routinely checked during these hours, will be recorded.

All the patients were administered 1000 mg iv paracetamol 30 minutes before the surgery ended, and was repeated every 6 hours following the surgery.The postoperative analgesia was evaluated by using VAS(Visual Analogue Scale).The PCA (Patient Controlled Analgesia) device was programmed at 10 μcq concentration with loading dose 50 μcq, 15-minute lock time, 25 μcq bolus without basal infusion, and this was continued for 24 hours in the postoperative recovery room.

ELIGIBILITY:
Inclusion Criteria:

* ASA (American Society of Anaesthesiologists) I-II-III group who will undergo liver resection surgery,
* no known history of heart, kidney, hematological disease, peptic ulcer, gastrointestinal bleeding, allergy, chronic pain
* who agreed to participate in the study

Exclusion Criteria:

* Patients with underlying serious cardiovascular disease,
* patients who cannot cooperate, patients who are allergic to one of the drugs to be used
* patients who do not want to participate

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2022-06-30 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-09-15 (Actual)

PRIMARY OUTCOMES:
Level of Pentraxin in ng/mL | After the Operation
  Pentraxin levels of the patients in both groups will be measured in terms ng/mL with Enzyme-Linked ImmunoSorbent Assay technique after the liver resection postoperatively.
Serum Amyloid A level in mcg/ml | After the operation
  Serum Amyloid A level of all patients in both groups will be measured in terms of mcg/ml with Enzyme-Linked ImmunoSorbent Assay technique after the liver resection postoperatively.

CONTACTS AND LOCATIONS:
Locations (1):
- Ataturk University, Erzurum, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Peralta C, Jimenez-Castro MB, Gracia-Sancho J. Hepatic ischemia and reperfusion injury: effects on the liver sinusoidal milieu. J Hepatol. 2013 Nov;59(5):1094-106. doi: 10.1016/j.jhep.2013.06.017. Epub 2013 Jun 25. PMID 23811302
- [Background] Siriussawakul A, Zaky A, Lang JD. Role of nitric oxide in hepatic ischemia-reperfusion injury. World J Gastroenterol. 2010 Dec 28;16(48):6079-86. doi: 10.3748/wjg.v16.i48.6079. PMID 21182222
- [Background] Ando T, Ito H, Kanbe A, Hara A, Seishima M. Deficiency of NALP3 Signaling Impairs Liver Regeneration After Partial Hepatectomy. Inflammation. 2017 Oct;40(5):1717-1725. doi: 10.1007/s10753-017-0613-6. PMID 28656530
- [Derived] Ates I, Laloglu E, Kara S, Yaman T, Isik B. The effects of dexmedetomidine and ketamine infusions on the inflammatory response in liver resection: A randomized double-blind placebo study. Medicine (Baltimore). 2025 Jul 4;104(27):e42999. doi: 10.1097/MD.0000000000042999. PMID 40629656